CLINICAL TRIAL: NCT04296942
Title: A Phase 1b Trial of Sequential Combinations of BN-Brachyury, Entinostat, Ado-trastuzuamb Emtansine and M7824 in Advanced Stage Breast Cancer (BrEAsT)
Brief Title: BN-Brachyury, Entinostat, Adotrastuzumab Emtansine and M7824 in Advanced Stage Breast Cancer (BrEAsT)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: One participant was accrued, and the study was stopped due to new safety data from the company for M7824 and slow accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fatima Karzai, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200056; 20-C-0056
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; HER2+ Breast Cancer; Hormone Receptor Negative Breast Cancer; Metastatic Breast Cancer
Keywords: Immuno-oncology; Immunotherapy; Vaccine; Invasive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — entinostat; bintrafusp alfa protein, human; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/M7824 (Bintrafusp alfa) + Bavarian Nordic (BN)-Brachyury (Experimental): Arm 1 - Triple Negative Breast Cancer.
  Bifunctional fusion molecule involving programmed death-ligand 1 (PD-L1) with transforming growth factor beta (TGF-b) sequestering agent added to a vaccine for the tumor associated antigen called brachyury.
  Interventions: Biological: Brachyury-TRICOM; Biological: M7824
- 2/M7824 + BN-Brachyury + Ado-trastuzumab emtansine (T-DM1) (Experimental): Arm 2 - Estrogen receptor (ER)-/progesterone receptor (PR)-/Human Epidermal Growth Factor Receptor 2 (HER2) + Breast Cancer.
  Bifunctional fusion molecule involving programmed death-ligand 1 (PD-L1) with transforming growth factor beta (TGF-b) sequestering agent added to a vaccine for the tumor associated antigen called brachyury. These investigational agents will be added to standard of care treatment called Ado-trastuzumab emtansine (T-DM1).
  Interventions: Biological: Brachyury-TRICOM; Biological: M7824; Biological: Ado-trastuzumab emtansine
- 3/M7824 + BN-Brachyury + T-DM1 + Entinostat (Experimental): Estrogen receptor (ER)-/progesterone receptor (PR)-/Human Epidermal Growth Factor Receptor 2 (HER2)+ Breast Cancer.
  Bifunctional fusion molecule involving programmed death-ligand 1 (PD-L1) with transforming growth factor beta (TGF-b) sequestering agent added to a vaccine for the tumor associated antigen called brachyury as well as to an oral histone deacetylase (HDAC) inhibitor called entinostat. These investigational agents will be added to standard of care treatment called Ado-trastuzumab emtansine (T-DM1). (T-DM1).
  Interventions: Biological: Brachyury-TRICOM; Drug: Entinostat; Biological: M7824; Biological: Ado-trastuzumab emtansine

INTERVENTIONS:
Biological: Brachyury-TRICOM — Every three weeks, until cycle 9, then every 12 weeks: *Recombinant MVA-Bavarian Nordic (BN)-Brachyury recommended phase 2 dose (R2PD): 4 injections of vaccines with 1 given subcutaneous (SC) in each extremity on Day 1 of Cycles 1 and 2. Each injection of MVA-BN-Brachyury consists of 2.0 x 10^8 infectious units (Inf.U). *Recombinant fowlpox virus (FPV)-BN-Brachyury: 1 injection given SC in one extremity on Day 1 of Cycles 3 and beyond. Each injection of FPV-BN-Brachyury consists of 1.0 x 10^9 Inf.U.
Drug: Entinostat — 5mg by mouth weekly (RP2D) administered by patient on Days 1, 8 and 15 of each cycle.
  Other Names: SNDX-275
  Arms: 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Biological: M7824 — 1800mg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
  Other Names: Bintrafusp alfa
Biological: Ado-trastuzumab emtansine — 3.6mg/kg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
  Other Names: T-DM1
  Arms: 2/M7824 + BN-Brachyury + Ado-trastuzumab emtansine (T-DM1); 3/M7824 + BN-Brachyury + T-DM1 + Entinostat

SUMMARY:
Background:

Breast cancer is the second most common cause of United States (U.S.) cancer deaths in women. Immunotherapy drugs use a person's immune system to fight cancer. Researchers want to see if a new combination of immunotherapy drugs can help treat breast cancer that has gone to places in the body outside of the breast (metastasized).

Objective:

To learn if a new combination of immunotherapy drugs can shrink tumors in people with metastatic breast cancer.

Eligibility:

Adults 18 and older who have been diagnosed with metastatic breast cancer, such as Triple Negative Breast Cancer (TNBC) or estrogen receptors (ER)-/progesterone receptors (PR)-/human epidermal growth factor receptor 2 (HER2)+ Breast Cancer (HER2+BC)

Design:

Participants will be screened with:

medical history

physical exam

disease confirmation (or tumor biopsy)

tumor scans (computed tomography, magnetic resonance imaging, and/or bone scan)

blood and urine tests

electrocardiogram (measures the hearts electrical activity)

echocardiogram (creates images of the heart).

Participants will be assigned to 1 of 3 groups. The drugs they get will be based on the group they are in. Drugs are given in cycles. Each cycle = 3 weeks. Participants will be seen in clinic every 3 weeks, prior to the start of a new cycle. At each visit, participants will have an clinical exam, have blood drawn and will be asked about any side effects. They will repeat the screening tests during the study. New scans, like a computed tomography (CT) scan, will be done every 6 weeks to see if the treatment is working.

All participants will get Bavarian Nordic (BN)-Brachyury. It is 2 different vaccines - a prime and a boost. First the priming vaccines, called MVA-BN-Brachyury help to jump start the immune system. Next the boosting vaccines, called fowlpox virus (FPV)-Brachyury help to keep the immune system going. They are injected under the skin during different cycles.

All participants will get M7824 (also known as Bintrafusp alfa), which is an immunotherapy drug. Some participants will get a commonly used drug is HER2+ breast cancer called adotrastuzumab emtansine (also known as T-DM1DM1 or kadcyla). For both, a needle is inserted into a vein to give the drugs slowly.

Some participants will take Entinostat weekly by mouth. It is in tablet form. Participants will keep a pill diary.

Participants will continue on their assigned treatment until their cancer grows, they develop side effects or want to stop treatment. About 28 days after treatment ends, participants will have a follow-up visit or a telephone call. Then they will be contacted every 3 months for 1 year, then every 6 months for 1 year. They may have more tumor scans or continue treatment.

DETAILED DESCRIPTION:
Background:

* Current greater than or equal to 2nd line treatments for metastatic breast cancer provide modest response rates, and modest improvement in progression-free survival but no treatments are curative.
* Bavarian-Nordic (BN)-Brachyury vaccine is a recombinant poxvirus vaccine against the transcription factor brachyury, which plays an important role in the epithelial-to-mesenchymal transition in breast cancer. A recently completed phase 1 study of BN-Brachyury vaccine showed the vaccine was well tolerated and generated an immune response.
* M7824 (Bintrafusp alfa) is a novel bifunctional fusion protein composed of a monoclonal antibody against human programmed death-ligand 1 (PD-L1) fused to the soluble extracellular domain of human transforming growth factor (TGF)-Beta receptor II (TGF-BetaRII(241-R2), which functions as a TGF-Beta trap.
* Ado-trastuzumab emtansine (T-DM1 or Kadcyla) is an antibody drug conjugate used in second- and third- line treatment of metastatic human epidermal growth factor receptor 2 (HER2+) breast cancer (HER2+BC). T-DM1 activates antibody-dependent cellular cytotoxicity (ADCC), dendritic cell maturation, increases tumor infiltrating lymphocytes (TILs), increased PD-L1 expression, and increased immunomodulatory cytokines.
* Entinostat is a class 1 histone deacetylase inhibitor (HDACi) which suppresses tumor initiating cells, regulatory T-cells and myeloid-derived suppressor cells (MDSCs), as well as enhances cytotoxic T-cell mediated lysis, direct natural killer (NK) lysis, NK cell activation, increases PD-L1 expression and antibody-dependent cellular cytotoxicity (ADCC). In addition, entinostat may also be able to overcome HER2 resistance.
* We propose a Phase 1b trial to evaluate the safety and efficacy of the stepwise combination of the BN-Brachyury vaccine, M7824, T-DM1 and entinostat in metastatic breast cancer.

  * Arm 1 - Triple Negative Breast Cancer (TNBC); M7824 + BN-Brachyury
  * Arm 2 - estrogen receptors (ER)-/progesterone receptors (PR-)/HER2+ Breast Cancer; M7824 + BN-Brachyury + T-DM1
  * Arm 3 - ER-/PR-/HER2+ Breast Cancer; M7824 + BN-Brachyury + T-DM1+ Entinostat

Objectives:

Primary Objectives:

* Arms 1-3: Overall response rate (overall response rate (ORR); partial response (PR)+complete response (CR)
* Arms 1-3: Safety for each of the three combinations of agents explored in the arms

Eligibility:

Selected Inclusion Criteria

* Histologically confirmed metastatic breast cancer with appropriate immunohistochemistry (IHC) testing by a certified lab:

  * For Arm 1: Triple negative breast cancer. Hormone receptor negative is defined by estrogen receptor < 10% and progesterone receptor < 10%. HER2 negative breast cancer is defined as HER2 per IHC 0 or 1+ or 2+ with negative fluorescence in situ hybridization (FISH).
  * For Arms 2 and 3: Hormone receptor negative, HER2+ breast cancer as defined by estrogen receptor < 10% and progesterone receptor < 10%. HER2 positive as per IHC 3+ or 2+ with positive FISH.
* Prior treatment:

  * For Arm 1: greater than or equal to 1 prior therapy in the metastatic setting. Patients with known PD-L1 positive tumors must have received prior treatment with atezolizumab + nab-paclitaxel. Patients with ER 1-9% must have received treatment with at least two lines of endocrine treatment (selective estrogen receptor modulators (SERM), AI, fulvestrant) with one prior treatment including a cyclin-dependent kinase 4 (CDK4)/6 inhibitor + endocrine therapy for their metastatic cancer and should be considered endocrine therapy resistant.
  * For Arms 2 and 3: greater than or equal to 1 prior treatment in the metastatic setting with a taxane (docetaxel or paclitaxel), herceptin and pertuzumab.
* Females or males greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Measurable metastatic disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* For Cohort 3, Arms 2 and 3: At least one biopsiable lesion and willingness to undergo up to three research biopsies.
* Adequate hematopoietic, hepatic, renal and cardiac (ejection fraction (EF) greater than or equal to 50%) function.

Selected Exclusion Criteria

* Patients who have received chemotherapy, including trastuzumab and pertuzumab in the previous 3 weeks; other investigational agents within 4 weeks or a programmed cell death protein 1 (PD-1)/PD-L1 antibody within 4 weeks prior to study enrollment; radiotherapy less than or equal to 4 weeks of study entry.
* Symptomatic central nervous system (CNS) metastases and leptomeningeal disease are excluded but treated brain metastases (no radiotherapy within 6 weeks) or asymptomatic brain metastasis are allowed.
* History of invasive malignancy less than or equal to 3 years prior to enrollment.
* History of congestive heart failure (CHF) as defined as New York Heart Association (NYHA) class 3 or 4 or hospitalization for CHF (any NYHA class) within 6 months of trial start.
* Concurrent use of chronic systemic steroids except for physiologic systemic steroids for replacement defined as 10mg of prednisone or an equivalent dose.

Design:

This study contains three separate, single arm phase 1b trials.

* Arm 1 will evaluate M7824 and BN-Brachyury in patients with triple-negative breast cancer (TNBC).
* If this doublet is determined to have acceptable toxicity (0-1 dose limiting toxicities (DLTs) of the first 6 patients), up to 19 patients will be enrolled on Arm 2 in which BN-Brachyury, M7824 and T-DM1 will be evaluated in patients with advanced HR-/HER2+ BC with disease progression after treatment with docetaxel (THP) or intolerance to THP.
* If this triplet is determined to have acceptable toxicity (0-1 DLTs of the first 6 patients), 19 patients will be enrolled on Arm 3 in which BN-Brachyury, entinostat, M7824 and T-DM1 will be evaluated in patients with advanced HR-/HER2+ BC with disease progression after treatment with THP or intolerance to THP.
* Up to 51 evaluable patients will be recruited for this study, with an accrual ceiling set at 65 patients.

Trial Drugs

* BN-Brachyury vaccine every 3 weeks until cycle 9, then every 12 weeks:

  * Recombinant MVA-BN-Brachyury (R2PD): 4 injections of vaccines with 1 given subcutaneous (SC) in each extremity on Day 1 of Cycles 1 and 2. Each injection of MVA-BN-Brachyury consists of 2.0 x 10(8) infectious units (Inf.U).
  * Recombinant fowlpox virus (FPV)-Brachyury: 1 injection given SC in one extremity on Day 1 of Cycles 3 and beyond. Each infection of FPV-Brachyury consists of 1.0 x 10(9) Inf.U.
* adotrastuzumab emtansine (T-DM1) 3.6mg/kg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
* M7824 2,400mg via IV infusion q3 weeks on Day 1 of each cycle.
* Entinostat 5mg by mouth weekly recommended phase 2 dose (RP2D) administered by patient on Days 1, 8 and 15 of each cycle.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed metastatic human epidermal growth factor receptor 2 (HER2+) breast cancer. HER2 positive or amplified breast cancer is defined as Immunohistochemistry (IHC) 3+ or fluorescence in situ hybridization (FISH) average HER2 copy number greater than or equal to 6 signals per cell or HER2/chromosome enumeration probe 17 (CEP17) greater than or equal to 2.0. HER2 testing must have been performed in a laboratory accredited by the College of American Pathology (CAP) or another accrediting entity.
* Patients must have hormone receptor negative, HER2+ breast cancer. Hormone receptor negative is defined as estrogen receptor < 10% by immunohistochemistry (IHC) and progesterone receptor < 10% by IHC.
* Patients must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patients must have at least one lesion deemed safe to biopsy and be willing to undergo up to three biopsies while on trial.
* Patients must have received front-line treatment for metastatic disease with a taxane, trastuzumab and pertuzumab (THP; docetaxel or paclitaxel allowed) and progressed on treatment or were intolerant to treatment. Patients must have received at least one prior therapy in the metastatic setting. Prior ado-trastuzumab (T-DM1) therapy is allowed.
* Female or male greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patients must have adequate bone marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL (> 1.5X 10(6)/L)
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin greater than or equal to 9 mg/dL (transfusion to obtain hemoglobin greater than or equal to 9 mg/dL within 24 hours prior to dosing is allowed)
* Patients must have adequate renal function, defined as:

  * serum creatinine less than or equal to 1.5 X upper limit of normal (ULN) OR
  * measured or calculated creatinine clearance greater than or equal to 60 mL/min for participant with creatinine levels > 1.5 X institutional ULN (Glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl).
* Patients must have adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than or equal to 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome, where bilirubin less than or equal to 5 mg/dL will be permitted. Gilbert's syndrome will be defined as elevated unconjugated bilirubin, with conjugated (direct) bilirubin within the normal range and less than 20% of the total. Total bilirubin will be permitted up to 5 mg/dL, if patients have historical readings consistent with the definition of Gilbert's syndrome prior to entering study. Adequate hepatic function for patients with known liver metastases is defined as AST and ALT levels less than or equal to 5 X ULN.
* Patients must have adequate cardiac function as defined by an ejection fraction greater than or equal to 50%.
* The effects of BN-Brachyury, entinostat, M7824 and T-DM1 on the developing human fetus are unknown. However, the two components of T-DM1 are known to have negative fetal effects including oligohydramnios and oligohydramnios sequence (pulmonary hypoplasia, skeletal malformations and neonatal death). For this reason:

  * Women of child-bearing potential must agree to use adequate contraception study entry, for the duration of study participation and for 7 months after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Men should refrain from fathering a child or donating sperm during the study and for 4 months after the last dose of study medications.
* Patients with well-controlled human immunodeficiency virus (HIV) infection are eligible for trial as long as:

  * On an effective anti-retroviral therapy (ART) 4 weeks and with evidence of viral suppression as defined as HIV viral load 400 copies/mL within the last 3 months;
  * Cluster of differentiation 4 (CD4) greater than or equal to 200 cells/microL within the last 3 months; and
  * No reported opportunistic infections within 6 months prior to enrollment, except for the following which will be allowed:

    i. Esophageal candidiasis treated within last 6 months or currently improving with antifungal treatment.

ii. Oral and/or genital herpes simplex virus (HSV) treated within last 6 months or currently improving with antiviral treatment.

iii. Mycobacterium avium infection in last 6 months or that has been treated for at least 1 month.

* Patients with evidence of chronic hepatitis B virus (HBV) infection are eligible for trial as long as the HBV viral load is undetectable on suppressive therapy, if indicated.
* Patients with history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable or unquantifiable HCV ribonucleic acid (RNA) 12 weeks or longer after definitive treatment completion.
* Patients must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have received chemotherapy, including herceptin and/or pertuzumab in the prior 3 weeks (6 weeks for nitrosoureas or mitomycin); other investigational agents or a programmed cell death protein 1/programmed death-ligand 1 (PD-1/L1) agent within 4 weeks prior to study enrollment.
* Patients who have received radiotherapy within 4 weeks prior to study entry.
* Patients with active brain metastases or leptomeningeal metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients with treated brain metastases are eligible if there is no magnetic resonance imaging (MRI) evidence of progression for 6 weeks after treatment is complete (no radiotherapy within 6 weeks) and within 28 days prior to the first dose of trial drug or asymptomatic brain metastasis. Patients requiring immunosuppressive doses of systemic corticosteroids (> 10mg/day prednisone equivalent) for palliation are excluded.
* Patients with a history of another invasive malignancy less than or equal to 3 years prior to enrollment (patients with non-melanoma skin cancers, carcinoma in situ of the breast or cervix are eligible).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study. For example, reaction to prior vaccination with vaccinia virus or known hypersensitivity reaction to fully humanized monoclonal antibodies (Grade greater than or equal to 3 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAEv5).
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection that requires systemic treatment with ongoing antibiotics (eligible if can stop antibiotics on day of enrollment), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that in the opinion of the primary investigator would prohibit the patient from complying with study requirements.
* Known history of a gastrointestinal illness that in the investigator's opinion would prevent the absorption of entinostat, which is an oral agent. (Arm 3 ONLY)
* Patients with bone metastases who have initiated denosumab or a bisphosphonate therapy within 28 days prior to or after Cycle 1 Day 1. Continuation of prior therapy is allowed.
* Patients with inherited bleeding disorders, a history of bleeding diathesis such as von Willebrand Factor (VWF) deficiency or recent (within 3 months prior to enrollment) clinically significant bleeding events that, in the judgment of the investigator, would interfere with patient's ability to carry out the treatment program.
* Patients should have no evidence of being immunocompromised as listed below:

  * Active, known or suspected autoimmune disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to an autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger in the opinion of the primary investigator.
  * Altered immune function, that in the judgement of the principal investigator (PI) that may affect a patient's ability to adequately engage the immune system and respond to the immunotherapy agents being administered, including but not limited to: inflammatory bowel disease; active infectious enteritis; eosinophilic enteritis; lupus erythematous; ankylosing spondylitis; scleroderma; multiple sclerosis. These criteria do not include all disease with an immune-related component but are not autoimmune in nature or have a primary alteration in the general immune function that may interfere with the vaccine mechanism of action, for example celiac disease.
  * Immunosuppressive therapy post-organ transplant.
* Concurrent use of chronic use of systemic steroids, except for physiologic doses of systemic steroids for replacement, defined as 10mg of prednisone per day or equivalent, or local (topical, nasal, ophthalmic or inhaled) steroid use or prior concomitant use with chemotherapy. Systemic steroids must have been discontinued >2 weeks prior to trial start. Prior use of corticosteroids in short-term schemes (duration shorter than 3 days) for indications such as prophylaxis of reactions to intravenous contrast for imaging studies or chemotherapy-related adverse events (AEs) are not considered part of this exclusion. Prior use of corticosteroids for brain metastasis ending at least 14 days prior to enrollment is not considered part of this exclusion criteria.
* Pregnant and breastfeeding women are excluded from this study because of the potential for teratogenic or abortifacient effects with all of the agents involved in this trial.
* Clinically significant cardiomyopathy, coronary disease, chronic heart failure (CHF; New York Heart Association class III or IV or hospitalization for CHF), or cerebrovascular accident within 6 months prior to enrollment.
* Patients with a history of myocarditis are excluded due to the potential of myocarditis with anti-PD-L1 antibodies.
* Patients with pulse oximetry < 92% on room air will be excluded due to the potential of pneumonitis with anti-PD-L1 antibodies.
* Any other condition, which would, in the opinion of the Principal Investigator or Medical Monitor, indicated the subject is a poor candidate for the clinical trial or would jeopardize the subject or the integrity of the data obtained.

ELIGIBILITY CRITERIA FOR ARMS 2 AND 3: M7824, BN-BRACHYURY, T-DM1 +/- ENTINOSTAT IN HER2+BC

INCLUSION CRITERIA:

* Patients must have histologically or cytologically confirmed metastatic HER2+ breast cancer. HER2 positive or amplified breast cancer is defined as IHC 3+ or FISH average HER2 copy number greater than or equal to 6 signals per cell or HER2/CEP17 greater than or equal to 2.0. (117) HER2 testing must have been performed in a laboratory accredited by the College of American Pathology (CAP) or another accrediting entity.
* Patients must have hormone receptor negative, HER2+ breast cancer. Hormone receptor negative is defined as estrogen receptor < 10% by IHC and progesterone receptor <10% by IHC.
* Patients must have measurable disease, per RECIST 1.1.
* Patients in Cohort 3 must have at least one lesion deemed safe to biopsy and be willing to undergo up to three biopsies while on trial.
* Patients must have received front-line treatment for metastatic disease with a taxane, trastuzumab and pertuzumab (THP; docetaxel or paclitaxel allowed) and progressed on treatment or were intolerant to treatment. Patients must have received at least one prior therapy in the metastatic setting. Prior T-DM1 therapy is allowed.
* Female or male greater than or equal to 18 years.
* ECOG performance status 0 or 1
* Patients must have adequate bone marrow function as defined below:

  * absolute neutrophil count greater than or equal to1,500/mcL (greater than or equal to 1.5X 106/L)
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin greater than or equal to 9 mg/dL (transfusion to obtain hemoglobin greater than or equal to 9 mg/dL within 24 hours prior to dosing is allowed)
* Patients must have adequate renal function, defined as:

  * serum creatinine less than or equal to 1.5 X upper limit of normal (ULN) OR
  * measured or calculated creatinine clearance greater than or equal to 60 mL/min for participant with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl).
* Patients must have adequate hepatic function, defined as AST and ALT levels less than or equal to 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome, where bilirubin less than or equal to 5 mg/dL will be permitted. Gilbert's syndrome will be defined as elevated unconjugated bilirubin, with conjugated (direct) bilirubin within the normal range and less than 20% of the total. Total bilirubin will be permitted up to 5 mg/dL, if patients have historical readings consistent with the definition of Gilbert's syndrome prior to entering study. Adequate hepatic function for patients with known liver metastases is defined as AST and ALT levels less than or equal to 5 X ULN.
* Patients must have adequate cardiac function as defined by an ejection fraction greater than or equal to 50%.
* The effects of BN-Brachyury, entinostat, M7824 and T-DM1 on the developing human fetus are unknown. However, the two components of T-DM1 are known to have negative fetal effects including oligohydramnios and oligohydramnios sequence (pulmonary hypoplasia, skeletal malformations and neonatal death). For this reason,

  * Women of child-bearing potential must agree to use adequate contraception study entry, for the duration of study participation and for 7 months after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fatima H Karzai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0056.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury: Arm 1 - Triple Negative Breast Cancer.
  Bifunctional fusion molecule involving programmed death-ligand 1 (PD-L1) with transforming growth factor beta (TGF-b) sequestering agent added to a vaccine for the tumor associated antigen called brachyury.
  Brachyury-TRICOM: Every three weeks, until cycle 9, then every 12 weeks: *Recombinant MVA-Bavarian Nordic (BN)-Brachyury recommended phase 2 dose (R2PD): 4 injections of vaccines with 1 given subcutaneous (SC) in each extremity on Day 1 of Cycles 1 and 2. Each injection of MVA-BN-Brachyury consists of 2.0 x 10^8 infectious units (Inf.U). *Recombinant fowlpox virus (FPV)-BN-Brachyury: 1 injection given SC in one extremity on Day 1 of Cycles 3 and beyond. Each injection of FPV-BN-Brachyury consists of 1.0 x 10^9 Inf.U.
  M7824: 1800mg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
- 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1): Arm 2 - Estrogen receptor (ER)-/progesterone receptor (PR)-/Human Epidermal Growth Factor Receptor 2 (HER2) + Breast Cancer.
  Bifunctional fusion molecule involving programmed death-ligand 1 (PD-L1) with transforming growth factor beta (TGF-b) sequestering agent added to a vaccine for the tumor associated antigen called brachyury. These investigational agents will be added to standard of care treatment called Ado-trastuzumab emtansine (T-DM1).
  Brachyury-TRICOM: Every three weeks, until cycle 9, then every 12 weeks: *Recombinant MVA-Bavarian Nordic (BN)-Brachyury recommended phase 2 dose (R2PD): 4 injections of vaccines with 1 given subcutaneous (SC) in each extremity on Day 1 of Cycles 1 and 2. Each injection of MVA-BN-Brachyury consists of 2.0 x 10^8 infectious units (Inf.U). *Recombinant fowlpox virus (FPV)-BN-Brachyury: 1 injection given SC in one extremity on Day 1 of Cycles 3 and beyond. Each injection of FPV-BN-Brachyury consists of 1.0 x 10^9 Inf.U.
  M7824: 1800mg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
  Ado-trastuzumab emtansine: 3.6mg/kg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
- 3/M7824 + BN-Brachyury + T-DM1 + Entinostat: Arm 3 - Estrogen receptor (ER)-/progesterone receptor (PR)-/Human Epidermal Growth Factor Receptor 2 (HER2)+ Breast Cancer.
  Bifunctional fusion molecule involving programmed death-ligand 1 (PD-L1) with transforming growth factor beta (TGF-b) sequestering agent added to a vaccine for the tumor associated antigen called brachyury as well as to an oral histone deacetylase (HDAC) inhibitor called entinostat. These investigational agents will be added to standard of care treatment called Ado-trastuzumab emtansine (T-DM1). (T-DM1).
  Brachyury-TRICOM: Every three weeks, until cycle 9, then every 12 weeks: *Recombinant MVA-Bavarian Nordic (BN)-Brachyury recommended phase 2 dose (R2PD): 4 injections of vaccines with 1 given subcutaneous (SC) in each extremity on Day 1 of Cycles 1 and 2. Each injection of MVA-BN-Brachyury consists of 2.0 x 10^8 infectious units (Inf.U). *Recombinant fowlpox virus (FPV)-BN-Brachyury: 1 injection given SC in one extremity on Day 1 of Cycles 3 and beyond. Each injection of FPV-BN-Brachyury consists of 1.0 x 10^9 Inf.U.
  Entinostat: 5mg by mouth weekly (RP2D) administered by patient on Days 1, 8 and 15 of each cycle.
  M7824: 1800mg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
  Ado-trastuzumab emtansine: 3.6mg/kg via intravenous (IV) infusion every (q)3 weeks on Day 1 of each cycle.
Period: Overall Study
Arm/Group | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Study closure by sponsor | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in group 2 and 3 due to study closure by the sponsor.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 1 |  |  | 1
  >=65 years | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (0) |  |  | 44.4 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 1 |  |  | 1
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 1 |  |  | 1
  White | 0 |  |  | 0
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (Partial Response + Complete Response) for Participants With Triple Negative Breast Cancer (TNBC)
Description: Overall response is defined as the best response (Partial Response + Complete Response) recorded from the start of treatment until disease progression/recurrence assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progression is at least a 20% increase in the sum of diameters of target lesions. appearance of new lesions. Appearance of one or more new lesions.
Time Frame: From start of treatment until disease progression/recurrence, approximately 5 months and 17 days.
Population: This outcome measure pertains to Arm 1 TNBC participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury
Number analyzed (Participants) | 1
Participants
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 1

2. Primary Outcome: Overall Response (Partial Response + Complete Response) for Participants With Human Epidermal Growth Factor Receptor 2 (HER2) + Breast Cancer (BC)
Description: Overall response is defined as the best response (Partial Response + Complete Response) recorded from the start of treatment until disease progression/recurrence. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progression is at least a 20% increase in the sum of diameters of target lesions. appearance of new lesions. Appearance of one or more new lesions.
Time Frame: From start of treatment until disease progression/recurrence, approximately 5 months and 17 days.
Population: This outcome measure pertains to Arm 2 and 3 only. Overall response in the HER2+ breast cancer cohort was not assessed as the study closed to accrual and no participants with HER2+ breast cancer was accrued.
Arm/Group | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants Experiencing at Least One Grade 3 to 5 Adverse Events for Each of the Three Combinations of Agents
Description: Adverse events were recorded using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 5 months and 17 days.
Population: No participants were enrolled in group 2 and 3 due to study closure by the sponsor.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Number analyzed (Participants) | 1 | 0 | 0
Participants
  Grade 3 | 0 |  |
  Grade 4 | 0 |  |
  Grade 5 | 0 |  |

4. Secondary Outcome: Progression-free Survival (PFS) in Triple Negative Breast Cancer (TNBC)
Description: Progression free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. In the absence of progression or death, PFS is censored at the date of last disease evaluation. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1 and is defined as at least a 20% increase in the sum of diameters of target lesions. appearance of new lesions. Appearance of one or more new lesions.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, approximately 5 months and 17 days.
Population: This outcome measure pertains to Arm 1 TNBC participants only.
Measure: Number; unit: Days
Arm/Group | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury
Number analyzed (Participants) | 1
Days | 63

5. Secondary Outcome: Progression Free Survival (PFS) in Participants With Metastatic Hormone Receptor (HR)-/Human Epidermal Growth Factor Receptor 2 (HER2) + Metastatic Breast Cancer Who Progressed on Initial Treatment With THP
Description: as for outcome 4
Time Frame: From start of treatment to time of progression or death, whichever occurs first, approximately 5 months and 17 days.
Population: This outcome measure pertains to Arm 2 and 3 only. PFS in the HER2+ breast cancer cohort was not assessed as the study closed to accrual and no participants with HER2+ breast cancer was accrued.
Arm/Group | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression Free Survival (PFS) in Participants With Metastatic Human Epidermal Growth Factor Receptor 2 (HER2+) Metastatic Breast Cancer Who Progressed on Initial Treatment With Docetaxel (THP)
Description: as for outcome 4
Time Frame: From start of treatment to time of progression or death, whichever occurs first, approximately 5 months and 17 days.
Population: as for outcome 5
Arm/Group | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Absolute Percentage of Stromal Tumor Infiltrating Lymphocytes (TILs) in Metastatic Deposits in Participants With Metastatic Human Epidermal Growth Factor Receptor 2 (HER2+) Metastatic Breast Cancer
Description: The absolute percentage of stromal TILs was measured by the Salgado method in metastatic deposits in participants with metastatic HER2+ metastatic breast cancer. The Salgado method is a standardized approach for measuring the percentage of stromal TILs in primary breast tumor specimens before therapy, using visual assessment of standard hematoxylin and eosin (H&E)-stained sections.
Time Frame: Baseline and on Cycle 3 Day 1
Population: This outcome measure pertains to Arm 2 and 3 only. No participants with HER2+ metastatic breast cancer was accrued and thus outcome measure is not possible to determine.
Arm/Group | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 5 months and 17 days.
Population: No participants were enrolled in group 2 and 3 due to study closure by the sponsor.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
Number analyzed (Participants) | 1 | 0 | 0
Participants | 1 |  |

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 5 months and 17 days.
Description: No participants were enrolled in group 2 and 3 due to study closure by the sponsor.
Arm/Group | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/M7824 (Bintrafusp Alfa) + Bavarian Nordic (BN)-Brachyury (N=1) | 2/M7824 + BN-Brachyury + Ado-trastuzumab Emtansine (T-DM1) (N=0) | 3/M7824 + BN-Brachyury + T-DM1 + Entinostat (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (3) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | NA
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04296942/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04296942/ICF_001.pdf